CLINICAL TRIAL: NCT04692246
Title: Effect of Essential Oils as Adjutants on the Treatment of Subjects With Periodontitis: Assessment of Metabolic Variables as Effect Modifiers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 Pandemic
Sponsor: Universidad de Granada (Other)
Collaborators: University of Palermo (Other)
Responsible Party: Principal Investigator, Francisco Mesa, Full Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PON-FSE-2017-1
Record Dates: First submitted 2020-12-22; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Periodontitis
Keywords: Anti-inflammation; Nutraceuticals; Periodontal therapy; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Patients that will receive the application of the extract in form of irrigation solutions in the periodontal pockets during regular periodontal treatment. Patients would continue at home during the follow-up period, taking the essential oils in as a rinse twice per day, and as a spray when regular toothbrush could not be performed.
  Interventions: Other: Plant-based oral rinse
- Control Group (Placebo Comparator): Patients that will follow the same protocol, but using placebo irrigation and a placebo spray at home.
  Interventions: Other: Placebo oral rinse

INTERVENTIONS:
Other: Plant-based oral rinse — Oral rinse enriched with plant-based essential oils.
  Arms: Test Group
Other: Placebo oral rinse — Oral rinse with the exact characteristics in terms of colour and odour of the plant-based one, but without the essential oils aimed to test in this study
  Arms: Control Group

SUMMARY:
Periodontitis, an infectious disease that affects the tooth-supporting tissues and shows a wide range of clinical, microbiological, and immunological manifestations, is associated with and probably caused by dynamic interaction among infectious agents, host immune responses, hazardous environmental exposure and genetic propensity. Bacteria are necessary for the disease to appear, but are not sufficient and do not account for all cases of periodontitis. According to one survey in the USA, chronic periodontitis affects approximately 46% of the adult population, with an even higher prevalence among the elderly. This prevalence refers to the cohort of young adults according to the WHO, with ages ranging from 35 to 44 years. Forms of periodontitis that appear at younger ages (before the age of 30 years), and that have other characteristics in addition to age, are known as aggressive periodontitis. The prevalence of this disorder ranges from 0.2% in Caucasians to 2.6% in Afro-Americans. The microbiota of the human oral mucosa together with other anatomical locations in the body constitute the human microbiome. The equilibrium between these organisms and the host response plays a fundamental role in human biology, both in health maintenance and in the appearance of disease. Unfavorable alterations in the composition of the microbiota are termed dysbiosis.

Antiseptics and antibiotics such as Chlorhexidine or Metronidazole, are delivered locally as an adjunct to scaling and root planing procedures, in order to eradicate the subgingival microbes, hence creating a healthy subgingival environment. However, the results presented in the literature are inconclusive. There is a need for further clinical trials with strict methodological criteria for allowing a more precise assessment of the efficacy of local antimicrobials in the treatment of chronic periodontitis.

Recently, there has been renewed interest in the application of natural products. Several natural products and herbs have claimed to have better properties and less side effects than chemical agents for irrigation. The use of natural extracts and essential oils as an irrigation agent for ultrasonic instrumentation has shown to promote slight adjunctive effect compared to chlorhexidine or water. In other study, natural extract showed a greater improvement compared to controls in patients with a more severe degree of periodontitis. However, in other studies this pocket reduction and clinical attachment gain were no significant when compared to water. Natural products have also been tested in forms of oral spray, and have shown to be effective against common oral pathogens without significant cytotoxicity in an in vitro study. Thus, it has the potential to prevent the infections and may serve as adjunctive treatment to conventional therapy. They claim to have the same or even more anti-microbial effect and anti-inflammatory effect without adding any chemicals. But still there is no adequate scientific evidence to support this hypothesis.

This study aims to test the effect as an adjutant to therapy of a nutraceutical composed of several plant extracts in patients with periodontitis and different levels of risk for metabolic syndrome. Specifically:

1. The response of periodontal clinical variables to non-surgical periodontal treatment in patients treated with the extract, compared to controls.
2. The effect on local inflammatory markers, in patients treated with the extract compared to controls.
3. The modifier effect of metabolic syndrome-related variables in the treatment outcomes of the patients treated with the extract compared to controls.

Hypothesis:

The application of the plant extract would act as an anti-inflammatory agent, contributing to better treatment outcomes of periodontitis, in terms of clinical and biochemical variables.

DETAILED DESCRIPTION:
METHODOLOGY

Study design Randomized, controlled, double-blinded clinical trial.

Study unit/population Subjects with diagnosis of periodontitis according to the joint EFP/AAP 2018 criteria for the case definition of periodontitis.

Inclusion criteria Patients attended in the University of Granada School of Dentistry (Granada, Spain) Signing of a written consent.

Exclusion criteria Age under 18 years, received periodontal treatment in the last year, anti-microbial therapy in the previous 3 months, multiple pregnancy and the presence of neoplastic or severe infectious diseases.

Sampling and randomization It is estimated to explore at least 60 patients, of which 30 will be randomized to each group, accordingly to similar studies on the topic available in the literature. The group allocation will also follow similar studies published previously in the field (7-9, 12, 13). All patients will receive standard periodontal treatment with an ultrasonic new generation device (AIRFLOW® Prophylaxis Master, EMS Dental, Nyon, Switzerland), and the group division will be based on the use of the extract as an adjunct to non-surgical treatment.

Test group: Patients that will receive the application of the extract in form of irrigation solutions in the periodontal pockets during regular periodontal treatment. Patients would continue at home during the follow-up period, taking the essential oils in as a rinse twice per day, and as a spray when regular toothbrush could not be performed.

Control group: Patients that will follow the same protocol, but using regular irrigation and a placebo spray at home.

The researchers that will perform the clinical examinations will be blinded for the group allocation of the participants, since the random allocation and prescription will be performed by a different researcher. Study products and placebo will be provided previously by the company BIONAP.

Study variables

1. Sociodemographic variables: sex, age, smoking habit (cigs/day), alcohol consumption (g/day).
2. Periodontal clinical variables:

   Periodontal examination will be performed by a calibrated researcher using PCPUNC15 periodontal probe (Hu-friedy, Chicago, IL, USA) and dental exploration mirror. Six surfaces in each implant will be measured: mesiovestibular, vestibular, distovestibular, distolingual, lingual, mesiolingual. All clinical data will be recorded in a periodontal chart. Clinical data will be gathered at baseline, and at 2 and 6 months of follow-up.

   Bleeding on probing: The percentage of bleeding implants while probing, will the registered following the index of Ainamo and Bay (14).

   Oral hygiene: Oral hygiene will be measured using the Plaque Index proposed by Tonetti (15). The presence of plaque will be registered by visual examination without using a plaque revealing agent.
3. Metabolic syndrome-related variables:

   * Body weight
   * Body height
   * Body mass index
   * Waist circumference
   * Blood pressure
4. Biochemical variables:

Samples of saliva, subgingival plaque and gingival crevicular fluid will be obtained at the beginning of the study, at 2 months and at the end of follow-up. A panel of inflammatory cytokines will be assessed.

Blood samples will be obtained at the beginning of the study, at 2 months and at the end of follow-up for the assessment of:

* Fasting blood glucose
* Lipid profile (Total cholesterol, Triglycerides, LDL-cholesterol and HDL-cholesterol).

Data management and statistical analysis A database in Excel format will be prepared including all recorded variables. The data will be analyzed by a single researcher. The statistical software SPSS v.21.0 (IBM Inc., Chicago, IL, USA) will be used, performing descriptive statistics (means, standard deviations and percentages) and analytical procedures (95% confidence intervals, Mann-Whitney test, Chi-square, Student's t-test for paired samples, and univariate and multivariate regression analysis). A 5% significance level will be considered for all tests.

ETHICAL CONSIDERATIONS The study will be designed in order to comply with the standards of the las revision of the Helsinki declaration. Approval from the Research Ethics Committee in Human Studies of the University of Granada will be obtained prior to the beginning of the study. Written informed consent will be obtained from all participants in the study. All obtained data will be anonymous and the study will be designed following the CONSORT guidelines for reporting clinical trials (16).

WORK PLAN

The project has been planned to be performed in a period of 2 years:

1. Study registration, ethical approval, and planning: December 2018 - February 2019.
2. Study enrollment, allocation, samples and data gathering. Follow-up period: March 2019 - April 2020.
3. Statistical analysis of all data: June 2020 - September 2020.
4. Manuscript preparation and publication process: October 2020 - April 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients attended in the University of Granada School of Dentistry (Granada, Spain)
* Accepting to be enrolled in the study and signing of a written consent.

Exclusion Criteria:

* Age under 18 years,
* Received periodontal treatment in the last year,
* Anti-microbial therapy in the previous 3 months
* Allergies
* Multiple pregnancy
* Presence of neoplastic or severe infectious diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | Change from Baseline Pocket probing depth at 3 months
  Depth of periodontal pockets present in the teeth of each patient in millimeters (mm) using a periodontal probe (PCPUNC-15)
Pocket probing depth | Change from Baseline Pocket probing depth at 6 months
  Depth of periodontal pockets present in the teeth of each patient in millimeters (mm) using a periodontal probe (PCPUNC-15)
Gingival recession | Change from Baseline Gingival recession at 3 months
  Distance from the gingival margin to the cemento-enamel junction in the teeth of each patient in millimeters (mm) using a periodontal probe (PCPUNC-15)
Gingival recession | Change from Baseline Gingival recession at 6 months
  Distance from the gingival margin to the cemento-enamel junction in the teeth of each patient in millimeters (mm) using a periodontal probe (PCPUNC-15)
Bleeding on probing | Change from Baseline Bleeding on probing at 3 months
  Percentage of teeth (%) that showed bleeding during periodontal examination.
Bleeding on probing | Change from Baseline Bleeding on probing at 6 months
  Percentage of teeth (%) that showed bleeding during periodontal examination.
Oral hygiene | Change from Baseline Visual Plaque Index at 3 months
  Percentage of teeth surfaces (4 in each tooth) that showed visible plaque during periodontal examination (Visual Plaque Index).
Oral hygiene | Change from Baseline Visual Plaque Index at 6 months
  Percentage of teeth surfaces (4 in each tooth) that showed visible plaque during periodontal examination (Visual Plaque Index).

SECONDARY OUTCOMES:
Body weight | Change from Baseline Body weight at 3 months
  Weight of each patient in kilograms (Kg) with a body scale.
Body weight | Change from Baseline Body weight at 6 months
  Weight of each patient in kilograms (Kg) with a body scale.
Body height | Baseline
  Height of each patient in centimeters (cm) with a scale.
Waist circumference | Change from Baseline Waist circumference at 3 months
  Waist abdominal circumference of each patient in centimeters (cm) with a measure tape.
Waist circumference | Change from Baseline Waist circumference at 6 months
  Waist abdominal circumference of each patient in centimeters (cm) with a measure tape.
Systolic Blood pressure | Change from Baseline Systolic Blood pressure at 3 months
  Systolic Blood pressure of each patient in Hg millimeters (Hg mm) measured with a sphygmomanometer.
Systolic Blood pressure | Change from Baseline Systolic Blood pressure at 6 months
  Systolic Blood pressure of each patient in Hg millimeters (Hg mm) measured with a sphygmomanometer.
Diastolic Blood pressure | Change from Baseline Diastolic Blood pressure at 3 months
  Diastolic Blood pressure of each patient in Hg millimeters (Hg mm) measured with a sphygmomanometer.
Diastolic Blood pressure | Change from Baseline Diastolic Blood pressure at 6 months
  Diastolic Blood pressure of each patient in Hg millimeters (Hg mm) measured with a sphygmomanometer.
Glycemia | Change from Baseline Glycemia at 3 months
  Fasting glycemia of each patient in milligrams per deciliter (mg/dL) measured with a glucometer.
Glycemia | Change from Baseline Glycemia at 6 months
  Fasting glycemia of each patient in milligrams per deciliter (mg/dL) measured with a glucometer.
Total cholesterol | Change from Baseline Total cholesterol at 6 months
  Total cholesterol levels of each patient in mg/dL measured in serum samples.
Triglyceride | Change from Baseline Triglyceride at 6 months
  Triglyceride levels of each patient in mg/dL measured in serum samples.
LDL-cholesterol | Change from Baseline LDL-cholesterol at 6 months
  Low-density lipoprotein levels of each patient in mg/dL measured in serum samples.
HDL-cholesterol | Change from Baseline HDL-cholesterol at 6 months
  High-density lipoprotein cholesterol levels of each patient in mg/dL measured in serum samples.

OTHER OUTCOMES:
Sex | Baseline
  Sex of the patient (male/female)
Age | Baseline
  Age of the patient at baseline examination
Smoking | Baseline
  Smoking habit of each patient in cigarrettes per day.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Mesa, PhD, Principal Investigator — Full Professor
Locations (1):
- University of Granada School of Dentistry, Granada, Spain

IPD SHARING:
Plan to Share IPD: No